CLINICAL TRIAL: NCT02002546
Title: Usefulness of a 2-hour Delta Troponin-I During the ED Identification and Exclusion of Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Chattanooga-Hamilton County Hospital Authority (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 13-069
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Heart Attack; Myocardial Infarction; Angina; Chest Pain
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina Pectoris; Chest Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED chest pain presenting patients

SUMMARY:
1. In chest pain patients with suspected acute coronary syndrome, a 2-hr delta Troponin-I as measured by the i-STAT immunoassay reliably identifies and excludes an acute myocardial infarction.
2. In chest pain patients with suspected acute coronary syndrome whose baseline troponin is above the 99th percentile but less than 0.2ng/ml, a 2hr delta Troponin-I as measured by the i-STAT immunoassay accurately discriminates between acute myocardial infarction and non-acute myocardial infarction troponin elevations.

DETAILED DESCRIPTION:
Primary Aims: 1) Demonstrate that a 2hr delta troponin as measured by the i-STAT platform can reliably identify and exclude MI on the initial ED evaluation. 2)Demonstrate that a 2hr delta troponin is useful in the discrimination AMI versus non-AMI conditions in patients with low abnormal baseline Troponin-I values.

Secondary Aims: 1) Demonstrate that a positive 2-hr delta troponin-I identifies patients at highest risk for 30 day ACE. 2) Other Secondary aims TBD.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years of age or older
2. Chest pain suspicious for ACS
3. Absence of ST-segment elevation AMI (STEMI) or STEMI equivalent on the initial ECG
4. Baseline i-STAT troponin less or equal to 1.0 ng/ml
5. Enrollment initiated before 2 hour 'delt' troponin value available for review
6. Ability and willingness to participate and cooperate with telephone follow-up evaluations

Exclusion Criteria:

1. ST-elevation or other ECG criteria that results in the diagnosis of AMI and results in patient being sent for percutaneous coronary interventions (PCI) or being treated with thrombolytics
2. Patients with chest pain not deemed to warrant cardiac screening
3. Blunt chest trauma
4. Tachyarrhythmia (ventricular tachycardia, supraventricular tachycardia, or rapid atrial fibrillation)
5. Cardiac Arrest prior to arrival
6. Hemodynamically unstable patients
7. Pulmonary edema requiring CPAP, BIPAP, or mechanical ventilation
8. Baseline i-STAT troponin measurement greater than 1.0 ng/ml
9. Baseline and 2-hour i-STAT Troponin measurements not obtained
10. Patient (or Legal Representative) unable or unwilling to provide written informed consent
11. Subject unwilling or unlikely to comply with study procedures, including protocol-specific blood sampling
12. Subject unwilling, unable, or deemed unlikely to respond or participate in telephone follow-up
13. Vulnerable populations as deemed inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the Emergency Department with chest pain or similar symptoms, and risk factors for ACS.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-09-04 (Actual)

PRIMARY OUTCOMES:
Change in Troponin value over a two hour interval. | 2 hours after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Erlanger Baroness Medical Center, Chattanooga, Tennessee, United States